CLINICAL TRIAL: NCT04441749
Title: TH-168: Needle Based Confocal Laser Endomicroscopy For The Diagnosis Of Peripheral Lung Nodules By Robotic Navigational Bronchoscopy
Brief Title: nCLE For Diagnosis Of Peripheral Lung Nodules By Robotic Navigational Bronchoscopy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Fox Chase Cancer Center (Other)
Collaborators: Mauna Kea Technologies (Industry); Johnson & Johnson (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-1006; TH-168 (Other: Fox Chase cancer Center)
Record Dates: First submitted 2020-06-15; First posted 2020-06-22 (Actual); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Diagnosis of Peripheral Lung Nodules

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tissue lung nodule) acquisition by transbronchial needle aspiration/ biopsy (standard of care)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- nCLE Analysis: Needle based confocal laser endomicroscopy (nCLE) employs a small fiber which can be passed through a biopsy needle to enable real time microscopic imaging of cells. With resolution of 3.5 microns it is possible to identify key features consistent with malignancy and pulmonary fibrosis
  Interventions: Device: Images acquired by needle-based Confocal Laser Endomicroscopy (nCLE)

INTERVENTIONS:
Device: Images acquired by needle-based Confocal Laser Endomicroscopy (nCLE) — Patients who are scheduled to undergo Robotic Navigational Bronchoscopy for a peripheral lung lesion will be enrolled. During bronchoscopy, confocal images will be captured using Cellvizio 100 Series Confocal Laser Imaging systems and their Confocal Miniprobes (Mauna Kea Technologies Paris, France). The Cellvizio system and miniprobes are FDA approved by 510(k) for use in through the respiratory tracts by endoscopy or endoscopic accessories. Only images and needle aspiration/ biopsy results from the expansion phase (20 patients) will be analyzed

SUMMARY:
Needle based confocal laser endomicroscopy (nCLE) employs a small fiber which can be passed through a biopsy needle to enable real time microscopic imaging of cells. With resolution of 3.5 microns it is possible to identify key features consistent with malignancy and pulmonary fibrosis. (Wijmans, et al., 2019). The effectiveness of nCLE with intravenous fluorescein has been demonstrated in central lung cancers using esophageal ultrasound guided needle placement (Wijmans, et al., 2019). In this study, the proposed nCLE lung cancer criteria had high accuracy for lung cancer detection and were consistently recognized by multiple raters. Probe based confocal microscopy (pCLE) has also been used in conjunction with a radial probe EBUS in evaluating solitary pulmonary nodules with a diagnostic accuracy of 79.2%. (Hassan, et al., 2017) Needle based confocal laser endomicroscopy (nCLE) has not previously been used in conjunction with robotic navigational bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Men and women, regardless of race, ethnic group or sexual orientation are eligible for this study.
* Patients undergoing robotic navigational bronchoscopy for evaluation of indeterminate lung nodules with largest dimension size of 8-30 mm
* Age > 18 years.
* Patients must have normal organ and marrow functions as defined below:

Leukocytes > 3,000/mcL Absolute neutrophil count > 1,500/mcL Total bilirubin within normal institutional limits Hemoglobin ≥7.0 AST/ALT (SGOT/SGPT) < 2 times institutional normal limits Creatinine OR Creatinine Clearance within normal institutional limits OR > 60 Ml/min/1.73 m2 for patients with creatinine levels above institutional normal

* Ability to understand and willingness to sign a written informed consent and HIPAA consent document
* WOCBP must agree not to get pregnant until after the day of the procedure

Exclusion Criteria:

* Patients with uncorrectable coagulopathy will be excluded.
* Known allergy to fluorescein or other contrast media
* Patients with hemodynamic instability will be excluded
* Patients with refractory hypoxemia will be excluded
* Patients with therapeutic anticoagulant that cannot be held for an appropriate interval prior to the procedure
* Patients who are unable to tolerate general anesthesia according to the anesthesiologist
* Patient requires chemotherapy
* Pregnant or breast feeding. Refer to section 4.5 for further detail.
* Subject has participated in an investigational drug or device research study within 30 days of enrollment that would interfere with this study
* Pregnancy:

Women of child-bearing potential (WOCBP) who are pregnant on the day of the procedure will be excluded from the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be enrolled from outpatient pulmonary clinic and from direct referrals from the inpatient pulmonary service and thoracic tumor board. Patients who scheduled to undergo Robotic Navigational Bronchoscopy for a peripheral lung lesion at Fox Chase Fox Center will be contacted to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-06-29 (Actual); Primary Completion 2021-09-20 (Actual); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Ability to obtain good quality nCLE images of lung nodules | 1 year
  Good quality nCLE images of lung nodules/ surrounding tissue in ≥80% of patients provided the peripheral lung nodule

CONTACTS AND LOCATIONS:
Locations (2):
- Fox Chase Cancer Center, Philadelphia, Pennsylvania, United States
- Amsterdam University Medical Center, Amsterdam, AZ, Netherlands

REFERENCES:
- [Derived] Manley CJ, Kramer T, Kumar R, Gong Y, Ehya H, Ross E, Bonta PI, Annema JT. Robotic bronchoscopic needle-based confocal laser endomicroscopy to diagnose peripheral lung nodules. Respirology. 2023 May;28(5):475-483. doi: 10.1111/resp.14438. Epub 2022 Dec 19. PMID 36535801